CLINICAL TRIAL: NCT05408481
Title: Hyponatremia in COVID-19 Patients With Adrenal Insufficiency and Its Relation to Mortality and Survival Scores.
Brief Title: Relation Between COVID-19 Pts and Hyponatremia in Adreno Ortical Insufficient Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Mostafa Abdel Raheem Gad El Rab, Dr, Assiut University
Other Study IDs: COVID-19 hyponatremia
Record Dates: First submitted 2022-06-04; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: Hyponatremia
MeSH Terms: conditions — COVID-19; Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum cortisol level — Biochemical test

SUMMARY:
Hyponatremia in COVID-19 patients with adrenal insufficiency

DETAILED DESCRIPTION:
Hyponatremia is the most prevalent hydroelectrolytic disorder in clinical practice, and is linked to higher rates of morbidity and mortality. 1, 2.Sodium balance disorder, particularly hyponatremia, is a common condition among hospitalized patients with COVID-19 . and it is associated with a higher risk of morbidity, mortality, and disability. Acute hyponatremia causes serious brain swelling that can lead to permanent disability or death. Chronic hyponatremia causes attention deficit, gait instability, and osteoporosis, Mechanisms of hyponatremia in coronavirus disease 2019 (COVID-19) patients. Osmotic syndrome of inappropriate antidiuretic hormone release (SIADH) as a major mechanism. Also hypovolemic hyponatremia that may have been common in COVID-19 patients since nausea, vomiting, diarrhea.we predict critical illness-related corticosteroid insufficiency (CIRCI) play a role in hyponatremia in COVID-19 , high percentage of critically ill patients with severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) infection in the study were treated with vasopressors (2). Angiotensin-converting enzyme 2 receptor and transmembrane serine protease 2 serine protease were colocalized in adrenocortical cells in the zona fasciculata and zona reticularis (2). plasma cortisol concentrations will be collected in critically ill patients with COVID-19 (2). The cortisol levels of critically ill patients with COVID-19 were low(2).We aimed to identify the previlence and mortality rate of hyponatremia in covid 19 patient with adrenal insufficiency . Our studies will present in Assiut hospital university on patients in isolation ward from October 2021 to October 2022.

ELIGIBILITY:
Inclusion Criteria:

* 1-Suspected COVID-19 patients come to isolation hospital in Assuit. 2-Hyponatremia. 3- Adrenal insufficiency

Exclusion Criteria:

* Non-cooperative patients

Ages: 19 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The effect of hyponatremia on mortality of COVID-19 patient with adrenal insufficiency | Baseline
  Na level will be measured in COVID-19 patients with adrenal insufficiency